CLINICAL TRIAL: NCT05705934
Title: Investigation of The Effects of Holistic Group Exercise Program on Muscle Thickness and Physical Performance in Older Adults With Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ondokuz Mayıs University (Other)
Collaborators: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Kübra Tuz, Lecturer, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-1268
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Participants in this group will receive holistic-based group exercise program. All evaluations in this group will be done in the form of before and after. The exercise program will be applied for 12 weeks, 3 days a week.
  Interventions: Other: Exercise
- Group 2 (No Intervention): Participants in this group will continue their routine habits and nutrition programs. All assessments in this group will be done in the form of before and after.

INTERVENTIONS:
Other: Exercise — Each session of the exercise program will last 50 minutes and will consist of 4 stages. At these stages, it is aimed to work the social, physical, spiritual and mental parameters of the holistic approach.
  Arms: Group 1

SUMMARY:
A decrease in muscle mass and function can cause the development of many chronic diseases, including sarcopenia. It has been reported that the best intervention for sarcopenia is exercise. Despite this, the optimal type of exercise for sarcopenia has not yet been determined. Although the holistic approach is used in the literature in the elderly population, it is noticeable that it does not find much space for itself in this patient group. In this study, it was aimed to examine the effects of holistic approach-based exercise program on individuals with sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 65
* Getting a diagnosis of sarcopenia
* To be able to walk at least 10 meters independently in public
* Getting a score of 4 and above from the clock drawing test
* Volunteer individuals

Exclusion Criteria:

* Having a neurological disease
* Having an uncontrollable cardiopulmonary disease
* Acute illness that will prevent him/her from understanding and performing the exercises to be performed status or the presence of significant cognitive impairment
* Providing continuity for less than 80% of the exercise program

Ages: 65 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-03-30 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Muscle Mass | Change from baseline at 12 weeks
  Muscle ultrasound (US) is a feasible and practical tool to predict sarcopenia. It provides scope for the efficient assessment of muscle quality whilst providing insight into the pathophysiology of sarcopenia in addition to the diagnosis of low muscle mass. US has distinct advantages over other available modalities for muscle mass because the tool allows for separate measurements of individual muscle groups in addition to being safe and portable.
The Timed Up&Go Test | Change from baseline at 12 weeks
  It is a balance test used in the evaluation of functional mobility in the elderly. In the timed up and go (TUG) test, subjects are asked to rise from a standard armchair, walk to a marker 3 m away, turn, walk back, and sit down again. The elapsed time in this sequence is recorded in seconds. Patients wear their regular footwear and can use a walking aid, if needed.
Short Physical Performance Battery (SPPB) | Change from baseline at 12 weeks
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance). A patient's score below 10 is the inclusion criterion for sarcopenia.

SECONDARY OUTCOMES:
SARC-F Questionnaire | Change from baseline at 12 weeks
  There are 5 SARC-F components: Strength, Assistance with walking, Rise from a chair, Climb stairs and Falls. The scores range from 0 to 10, with 0 to 2 points for each component. A score equal to or greater than 4 is predictive of sarcopenia and poor outcome.
Charlson Comorbidity Index | Change from baseline at 12 weeks
  The Charlson Comorbidity Index is a method of categorizing comorbidities of patients based on the International Classification of Diseases (ICD) diagnosis codes found in administrative data. Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use.
30-Second Chair Stand Test | Change from baseline at 12 weeks
  The 30 Second Sit to Stand Test is also known as 30 second chair stand test ( 30CST), is for testing leg strength and endurance in older adults. In the middle part of the chair, the person's back is upright, his feet are pressed to the floor and his arms it is ensured that he sits diagonally in front of his chest (right hand on the left shoulder, left hand on the right shoulder). While the person is in this position, he starts the test with the start command and does it as fully as he can for 30 seconds he takes off; the exact number of departures he has made during 30 seconds constitutes the person's score. Scores less than 10 indicate poor muscle endurance.
Hand Grip Strength | Change from baseline at 12 weeks
  It is a method that provides reliable information about upper extremity muscle strength. Grip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles. It can be used as a screening tool for the measurement of upper body strength and overall strength. It is most useful when multiple measurements are taken over time to track performance.
Berg Balance Test | Change from baseline at 12 weeks
  The BBS consists of 14 different items that evaluate sitting, standing, and dynamic balance in a hierarchical manner and are assigned scores of 0 to 4, with 0 indicating that an individual is unable to complete the task entirely. The BBS comprises the following tasks: sit to stand; standing without support; sitting without support; stand to sit; transfers; standing with eyes closed; the Romberg test with eyes open; functional reach in standing; picking up something off the floor; turning and looking behind; a 360° turn to the right and left; toe touches to a stool; the sharpened Romberg test; and single-leg stance. A high score indicates good balance.
Depression | Change from baseline at 12 weeks
  The 15-item geriatric depression scale (GDS-15) is a short form of GDS and is used to screen, diagnose, and evaluate depression in elderly individuals. The cut-off point of the scale is 7 points and above.
Mini Nutritional Assessment (MNA) | Change from baseline at 12 weeks
  The Mini Nutritional Assessment (MNA) has recently been designed and validated to provide a single, rapid assessment of nutritional status in elderly patients in outpatient clinics, hospitals, and nursing homes. The MNA test is composed of simple measurements and brief questions that can be completed in about 10 min. In the test with a total score of 30, below 17 points is considered as significant malnutrition.